# Informed Consent Diagnostic Accuracy of the Water-Immersion Wrinkle Test for the Diagnosis of Small-Fiber Neuropathy

Principal Investigator: Dr. Lucas A. Piedrafita Vico – Hospital Británico de Buenos Aires.

NCT – pending assignment

October 9, 2024

By means of this document, we invite you to authorize us to collect information from your medical record, to perform the water-immersion wrinkle test, and to take photographs of the fingertips of your hands, given that you have been diagnosed with small-fiber neuropathy. This type of neuropathy may be characterized by sensory symptoms (loss or reduction of perception of cold and/or heat, altered nociceptive sensation [pain]) and may be accompanied by unpleasant symptoms (paresthesias such as tingling, pins and needles, burning).

# **Description of the Research Study**

Based on your medical history, we will transcribe your clinical data and the results of your tests using only a code that includes the initials of your name and your date of birth. This neuropathy poses diagnostic challenges due to the complexity of its manifestations and the currently available diagnostic tests. The water-immersion wrinkle test (WIWT) is a simpler, noninvasive, painless, and accessible tool that has the potential to make a valuable contribution to the initial diagnosis of your neuropathy, supporting the final diagnosis. The test involves immersing both hands in warm water (at 44-43°C) for 15 minutes and then observing the wrinkles that form on your fingertips; these provide information about the fibers affected in your neuropathy. We plan to compare this test with other tests that you have undergone because they are the traditional diagnostic methods for your neuropathy (such as quantitative sensory testing [QST], nerve conduction studies, and the sudomotor sympathetic response [SSR]) in order to assess the future usefulness of WIWT and help improve the comprehensive diagnosis of your neuropathy.

#### **Potential Benefits**

You will not receive any direct benefit for authorizing the collection of your health data and for undergoing the water-immersion wrinkle test; however, it is expected that this information will allow us to better understand the usefulness of the test and thereby improve the initial diagnosis of patients with small-fiber neuropathy. You are not expected to experience any risk or harm from allowing access to your data and undergoing this test. The treatment you receive for your condition will not be affected in any way.

#### Will my participation in the study be kept confidential?

All personal information we collect will be kept confidential on a computer accessible only to the physicians responsible for this study from the Department of Neurology at Hospital Británico de Buenos Aires. This database will be maintained in strict confidentiality and may only be viewed by the study investigators and by the Ethics Committee authorities, in accordance with the Personal Data Protection Law (Habeas Data Law No. 25.326). Your name will not be disclosed in any report or publication; instead, you will be identified by your initials and date of birth. The data and results of this study may also be presented at scientific meetings or in publications, but in such presentations the identities of the individuals participating in the study

will be kept confidential. By signing this form, you or your legal representative authorize such access.

#### **Communication of Results – New Information**

You may contact Dr. Lucas Piedrafita Vico (11-5958-8888) from the research team and Ms. Luciana Casella (43096892 – Institutional Review Board) at any time to obtain information about the progress of the study or its general results. You will be informed of any relevant data or new information that arises during the course of the study and that may be of diagnostic or therapeutic interest to you.

# Withdrawal from the Study

You may withdraw from this study at any time without this affecting your subsequent medical care.

#### Costs

Participation in this study will not entail any expenses of any kind for you.

# **Voluntary Participation**

Your participation is entirely free and voluntary. Your decision will not affect the quality of the health services you receive. You may take time to reflect and discuss your participation with peers or family members before giving us an answer. You are also free to withdraw from the research project at any time.

If you have questions about your rights or ethical issues related to your participation in this research study, you may contact the Ethics Committee of this hospital (Ms. Luciana Casella, phone 43096892) or the investigator. You are also informed that you may be selected by the Institutional Review Board (Comité de Revisión Institucional) to be interviewed regarding your understanding of and agreement with the study. Thank you for reading this document. We are at your disposal to answer any questions you may have.

### **Investigators**

Dr. Lucas Piedrafita Vico: 11-5958-8888

Email: lpiedrafita@hbritanico.com.ar

| <b>Informed Consent Declara</b> | tion | |
|---|---|---|
| patient or responsible family<br>informed consent form. I u<br>answered. I understand that<br>the health professionals at I<br>medical record, to perform<br>fingertips of my hands. All | member), confirm that I had not make the information properties I will receive a copy of this Hospital Británico de Bueno the water-immersion wrink of the above is related to evaluate. | (full name of the ave read—or have had read to me—this presented and my questions have been form. I voluntarily consent to authorize as Aires to collect information from my the test, and to take photographs of the raluating the usefulness of the test under it may be used in future studies. |
| Preservation of Informatio | n and Anonymous Photogr | aphs |
| [ ] I accept / [ ] I refuse that this study has ended. | at my information and photog | graphs be used in other research after |
| By signing this consent, I am<br>the hospital from their civil of | | s, nor am I releasing the investigator or |
| Patient's Signature | Printed Name and ID | Date of Signature |
| and that I have complied wit | h the Declaration of Helsinki<br>quired by the Institutional Re<br>lluated and approved this stud | This study to the above-named patient, i of the World Medical Association and eview Board of Hospital Británico de day and will verify compliance with all |